CLINICAL TRIAL: NCT05859568
Title: Baseline Performance and Fitting Parameters for Sonova Products
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Bionics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPR2301
Record Dates: First submitted 2023-05-05; First posted 2023-05-16 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Hearing Loss; Ear Diseases; Hearing Disorders; Otolaryngological Disease
MeSH Terms: conditions — Hearing Loss; Ear Diseases; Hearing Disorders; Otorhinolaryngologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Microphone Location versus Microphone Algorithm Comparison (Experimental): Comparing performance and subjective feedback for pinna-located microphone versus a pinna-simulated microphone algorithm.
  Interventions: Device: Pinna-located microphone; Device: Pinna-simulated microphone algorithm

INTERVENTIONS:
Device: Pinna-located microphone — Sound processors using a pinna-located microphone
Device: Pinna-simulated microphone algorithm — Sound processors using a pinna-simulated algorithm

SUMMARY:
The purpose of this study is to assess the effectiveness and optimization of various FDA approved products.

DETAILED DESCRIPTION:
This study uses a prospective within-subjects repeated-measures design in which each subject serves as her/his own control. The purpose of this study is to assess the effectiveness and optimization of various FDA approved hardware, signal preprocessing and processing software, fitting characteristics, and service delivery methods, such as remote support and/or tele-audiology on an expanded subject demographic. The insights gained from this study will be used to optimize listening configuration recommendations, refine audiological practice, and inform future innovations.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide Informed Consent/Assent
* Adults (age +18 years) and children (8-17 years) can be enrolled in this study

  * If child is aged 8-17 years, an assent will be completed, and the subject must be accompanied by a parent or legal guardian for all study activities
* Have the functional capability to operate the controls for the device and to comply with all directions during the study as determined by the investigator conducting the consent/baseline visit
* English language proficiency as determined by the investigator

Exclusion Criteria:

• Have any significant medical condition that, in the opinion of any of the investigators, is likely to interfere with study procedures or likely to confound evaluation of study endpoints

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2028-04-17 (Estimated); Study Completion 2028-04-17 (Estimated)

PRIMARY OUTCOMES:
Speech performance in noise | 1 day
  The primary efficacy endpoint is recorded AzBio sentences presented from a single loud speaker at 60 dBA. The recognition scores using the pinna-located microphone in quiet and noise captured at initial visit will be compared to the AzBio sentence recognition scores using the pinna-simulated microphone. Scores are determined on a scale of 0% to 100% words correct with higher scores indicating a better outcome.

SECONDARY OUTCOMES:
Localization performance | 1 day
  A secondary efficacy endpoint is a front/back localization task where filtered pink noise is presented at 60dBA from one of six speakers in a 360 degree array. Scores are generated in percent correct; the scores obtained from the pinna-located microphone will be compared to the localization scores using the pinna-simulated microphone.
Analysis of usability and preference questionnaire | 8 weeks
  Subject responses captured on a usability and preference questionnaire at the initial visit will be compared to responses on the questionnaire administered after each two-week chronic use interval. Questions will inquire about subject's ability and experience hearing and listening in different situations and wearing configuration preferences. The questions are rated on a 5-point Likert scale with varying strength, such as "It was easy to verify proper microphone function" with answers ranging from strongly disagree to strongly agree.

CONTACTS AND LOCATIONS:
Locations (1):
- Advanced Bionics, Valencia, California, United States

IPD SHARING:
Plan to Share IPD: No